CLINICAL TRIAL: NCT02692196
Title: Voluntary Regulation of Fronto-limbic Functional Connectivity: A Proof-of-concept Real-time fMRI Study
Brief Title: Fronto-limbic Functional Connectivity Via Real-time fMRI Neurofeedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Prof., University of Electronic Science and Technology of China
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-09
Record Dates: First submitted 2016-02-17; First posted 2016-02-25 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Healthy
Keywords: Neurofeedback; Emotion processing; Real-time; fMRI

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Neurofeedback Training (Experimental): Neurofeedback training - neurofeedback of fronto-limbic functional connectivity.
  Interventions: Device: Real-time fMRI neurofeedback from Turbo Brain voyager (TBV) 3.2
- Sham Control (Sham Comparator): Sham training - feedback that is not related with fronts-limbic connectivity (motor connectivity)
  Interventions: Device: Real-time fMRI neurofeedback from Turbo Brain voyager (TBV) 3.2

INTERVENTIONS:
Device: Real-time fMRI neurofeedback from Turbo Brain voyager (TBV) 3.2

SUMMARY:
Real-time fMRI neurofeedback training induced volitional control of brain activity and connectivity could help individuals to gain better control over their emotions.

DETAILED DESCRIPTION:
In the present proof-of-concept study, investigators plan to evaluate whether real-time fMRI neurofeedback training can enable individuals to gain volitional control over their fronto-limbic circuitry. Given that this circuitry has been abundantly implicated in emotional perception and regulation this could facilitate emotional control. Suitable participants underwent fronto-limbic connectivity feedback training and sham training in a cross over design. During both trainings participants are instructed to regulate the neural indices during feedback. We expect that receiving fronto-limbic feedback enhances emotion regulation during the training.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects without past or current psychiatric or neurological disorders

Exclusion Criteria:

* pregnant, taking oral contraceptives

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Neural indices of training success | three days
Training-induced changes in emotion related processing | three days
  The scores of visual analogue scale assessing individuals' anxiety level will be compared between before and after training within each group as well as between twe groups after training

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Becker, Dr., Principal Investigator — School of Life Science and Technology, University of Electronic Science and Technology of China
Locations (1):
- School of Life Science and Technology, University of Electronic Science and Technology of China, Chengdu, Sichuan, China